CLINICAL TRIAL: NCT06937346
Title: Robotic-Assisted Upper Limb Rehabilitation After Stroke Using the ReHand System: A Randomized Controlled Trial
Brief Title: Rehabilitation Robotic System ReHand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaganda Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2025-03-29; First posted 2025-04-22 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Rehabilitation; Robotic Exoskeleton
Keywords: Exoskeleton of the hand; rehabilitation; robotic system; recovery; cerebral stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group: Robot Rehand + Standard Rehabilitation (Experimental): The patients in the main group will undergo standard rehabilitation combined with the use of the ReHand robotic device, five times per week for 60 days.
  Interventions: Device: The Rehand Robotic Glove; Other: Standard Rehabilitation
- Control group: Standard Rehabilitation Only (Active Comparator): Patients in the control group will undergo standard rehabilitation, without the use of the ReHand robotic device. They will attend sessions 5 times per week for 60 days.
  Interventions: Other: Standard Rehabilitation

INTERVENTIONS:
Device: The Rehand Robotic Glove — The exoskeleton hand system provides recovery and training for paralyzed fingers using an innovative method that mirrors the movements of a healthy hand. The system uses a sensor glove to read movements and transfer them to a rehabilitation glove. This forces the injured hand to repeat the same movements as the healthy hand, helping to restore motor skills.
  The system combines flexible robotics with neuroscience to help patients retrain their muscles. It reduces muscle tension and swelling, relieves stiffness, improves blood circulation, and restores muscle performance after atrophy. It also reduces hypertension and joint pain, and activates neuroplasticity through passive and active techniques.
  All patients received standard rehabilitation treatments in accordance with clinical protocol No. 94 for the third stage of medical rehabilitation, approved by the Joint Commission on Quality of Medical Services from the Ministry of Health of Kazakhstan on 14 May 2020.
  Arms: intervention group: Robot Rehand + Standard Rehabilitation
Other: Standard Rehabilitation — All patients received standard rehabilitation treatments in accordance with clinical protocol No. 94 for the third stage of medical rehabilitation, approved by the Joint Commission on Quality of Medical Services from the Ministry of Health of Kazakhstan on 14 May 2020.

SUMMARY:
The aim of this clinical trial is to investigate the efficacy of the ReHand rehabilitation system for the recovery of patients after a stroke.

The main objectives of the study:

1. To assess the functional state of patients with cerebral stroke according to the The Barthel Index, on the Functional Independence Measure (FIM) scale of functional independence.
2. To assess the neurological deficit of patients according to the National Institutes of Health Stroke Scale (NIHSS), the state of function of the affected arm and the degree of fine motor impairment according to the The Frenchay Arm Test (FAT), The Fugl-Meyer Assessment for upper extremity (FMA-UE) scale, modified Wolf Motor Function Test (mWMFT), according to the upper limb disability questionnaire The Disabilities of the Arm, Shoulder, and Hand (DASH) test.
3. To investigate the state of psycho-emotional status in patients on the Hospital Anxiety and Depression Scale (HADS) of anxiety and depression.
4. To determine the effectiveness of the rehabilitation performed in patients with cerebral stroke after recovery by the ReHand system according to the above scales.

Participants:

All patients received standard rehabilitation methods according to the clinical protocol for diagnosis and treatment No. 94, "The third stage of medical rehabilitation", approved by the Joint Commission on the Quality of Medical Services of the Ministry of Health of the Republic of Kazakhstan on May 14, 2020.

The main group of patients underwent rehabilitation using a robotic glove for 8 weeks, with 5 classes per week and each class lasting 45 minutes.

The control group did not receive robotic glove-based rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* a stroke that occurred no more than six months prior;
* absence of somatic conditions that would interfere with the use of the hand exoskeleton system (such as rheumatoid arthritis, severe muscle hypertonia, joint pathology, fractures, etc.);
* clear consciousness;
* presence of upper limb and fine motor impairments;
* no history of recurrent cerebral strokes;
* no comorbidities associated with cognitive dysfunction (such as Parkinson's disease, Wernicke's encephalopathy, alcoholic encephalopathy, etc.) that would hinder instruction comprehension;
* absence of rheumatological issues (including contractures and significant pain syndromes) that would impede study participation;
* absence of acute or chronic (in the decompensated stage) diseases of internal organs;
* signing of informed consent for study participation;
* all participants were adults

Exclusion criteria:

* lack of clear consciousness,
* a history of recurrent cerebral stroke,
* a stroke that occurred more than 6 months ago,
* lack of upper limb function or fine motor disorders,
* the presence of concomitant diseases associated with cognitive dysfunction (such as Parkinson's disease, Wernicke encephalopathy, alcoholic encephalopathy, etc.) that may interfere with understanding the instructions,
* rheumatological diseases.
* problems (including contractures and severe pain syndromes) that could interfere with participation in the study,
* the presence of acute or chronic (decompensation stage) diseases of internal organs,
* contraindications according to Clinical Protocol No. 94 on diagnosis and treatment "The third stage of medical rehabilitation", approved by the Ministry of Health of the Republic of Kazakhstan on May 14, 2020 (frequent or severe bleeding of various origins; febrile or subfebrile fever of unknown origin; acute infectious diseases; acute osteomyelitis; acute deep vein thrombosis; complicated cardiac arrhythmias, heart failure in the active stage; active forms of tuberculosis; malignant tumors (IV clinical group).; respiratory failure of stage III and above; various purulent (pulmonary) diseases with significant intoxication; decompensated diseases such as irreversible metabolic disorders (diabetes mellitus, myxedema, thyrotoxicosis, etc.), functional insufficiency of the liver or pancreas of stage III; epilepsy in the seizure phase; mental disorders causing desocialization and emotional or behavioral disorders.; purulent skin diseases, infectious skin diseases (scabies, fungal infections, etc.); anemia with an Hb level of 90 g/l or lower;
* lack of signed informed consent to participate in the study.;
* he underage age of the participants.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Karaganda region, Karaganda, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amirbekova M, Kispayeva T, Izbassarova A, Adomaviciene A, Sorokina M, Zhunussova T. Rehabilitation of patients in the subacute phase of stroke using the ReHand robotic system: a randomized controlled trial. Front Hum Neurosci. 2025 Nov 24;19:1690643. doi: 10.3389/fnhum.2025.1690643. eCollection 2025. PMID 41377192

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 120 participants provided informed consent and were enrolled in the study. All enrolled participants were randomized into two groups, with 60 participants in each group.
Groups:
- Intervention Group: Robot Rehand + Standard Rehabilitation: The patients in the main group will undergo standard rehabilitation combined with the use of the ReHand robotic device, five times per week for 60 days.
  The Rehand Robotic Glove: The exoskeleton hand system provides recovery and training for paralyzed fingers using an innovative method that mirrors the movements of a healthy hand. The system uses a sensor glove to read movements and transfer them to a rehabilitation glove. This forces the injured hand to repeat the same movements as the healthy hand, helping to restore motor skills.
  The system combines flexible robotics with neuroscience to help patients retrain their muscles. It reduces muscle tension and swelling, relieves stiffness, improves blood circulation, and restores muscle performance after atrophy. It also reduces hypertension and joint pain, and activates neuroplasticity through passive and active techniques.
  All patients received standard rehabilitation treatments in accordance with clinical protocol No. 94 for the third stage of medical rehabilitation, approved by the Joint Commission on Quality of Medical Services from the Ministry of Health of Kazakhstan on 14 May 2020.
  Standard Rehabilitation: All patients received standard rehabilitation treatments in accordance with clinical protocol No. 94 for the third stage of medical rehabilitation, approved by the Joint Commission on Quality of Medical Services from the Ministry of Health of Kazakhstan on 14 May 2020.
Period: Overall Study
Arm/Group | Intervention Group: Robot Rehand + Standard Rehabilitation | Control Group: Standard Rehabilitation Only
Started | 60 (All randomized participants (60 in the experimental group) started the assigned intervention.) | 60 (All randomized participants ( 60 in the control group) started the assigned intervention.)
Completed | 60 (All randomized participants (60 per group) completed the intervention and the final assessment (Day 60). No major protocol deviations occurred.) | 60 (All randomized participants (60 per group) completed the intervention and the final assessment (Day 60). No major protocol deviations occurred.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group: Robot Rehand + Standard Rehabilitation | Control Group: Standard Rehabilitation Only | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (9.0) | 59.3 (10.0) | 59.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 46 | 44 | 90
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Type of stroke [Count of Participants; unit: Participants]
  Ischemic | 44 | 45 | 89
  Hemorrhagic | 16 | 15 | 31
Days after stroke [Mean (Standard Deviation); unit: days] | 104.2 (45.0) | 106.0 (46.7) | 105.1 (45.6)
Fugl-Meyer Assessment for Upper Extremity (FMA-UE) [Median (Inter-Quartile Range); unit: score on a scale] — Fugl-Meyer Assessment for Upper Extremity; range: 0-66 points; higher scores indicate better motor function and less impairment.
  score on a scale | 29.0 [24.8 to 32.0] | 29.0 [26.0 to 32.0] | 29.0 [25.8 to 32.0]
Barthel Index (BI) [Median (Inter-Quartile Range); unit: score on a scale] — Barthel Index; range: 0-100 points; higher scores indicate greater independence in activities of daily living.
  score on a scale | 40.0 [35.0 to 40.0] | 45.0 [40.0 to 50.0] | 40.0 [40.0 to 45.0]
National Institutes of Health Stroke Scale(NIHSS) [Median (Inter-Quartile Range); unit: score on a scale] — National Institutes of Health Stroke Scale (NIHSS); range: 0-42 points; higher scores indicate more severe neurological impairment.
  score on a scale | 8.0 [7.0 to 11.0] | 8.0 [5.8 to 11.0] | 8.0 [6.0 to 11.0]
Functional Independence Measure (FIM) [Median (Inter-Quartile Range); unit: score on a scale] — Functional Independence Measure (FIM); range: 18-126 points; higher scores indicate greater functional independence.
  score on a scale | 52.0 [50.0 to 55.2] | 54.5 [52.0 to 58.0] | 54.0 [50.0 to 57.0]
Frenchay Arm Test (FAT) [Median (Inter-Quartile Range); unit: score on a scale] — Frenchay Arm Test (FAT); range: 0-5 points; higher scores indicate better arm function.
  score on a scale | 1.0 [0.0 to 1.0] | 1.0 [0.0 to 1.0] | 1.0 [0.0 to 1.0]
modified Wolf Motor Function Test (mWMFT) [Median (Inter-Quartile Range); unit: score on a scale] — modified Wolf Motor Function Test (mWMFT) total score range: 0-75 points; higher scores indicate better upper extremity motor function.
  score on a scale | 36.0 [33.0 to 39.0] | 37.0 [34.0 to 40.0] | 36.5 [33.8 to 39.2]
Disabilities of the Arm, Shoulder and Hand (DASH) [Median (Inter-Quartile Range); unit: score on a scale] — Disabilities of the Arm, Shoulder and Hand (DASH); range: 0-100 points; higher scores indicate greater disability.
  score on a scale | 46.0 [43.0 to 48.0] | 46.5 [44.0 to 49.2] | 46.0 [43.0 to 49.0]
Hospital Anxiety and Depression Scale (HADS) [Median (Inter-Quartile Range); unit: score on a scale] — Hospital Anxiety and Depression Scale (HADS); range: 0-42 points; higher scores indicate greater psychological distress (more severe anxiety and depression symptoms).
  score on a scale | 28.0 [25.0 to 33.0] | 31.0 [28.0 to 34.0] | 30.0 [26.8 to 33.2]

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment for Upper Extremity (FMA-UE)
Description: Fugl-Meyer Assessment for Upper Extremity (FMA-UE); range: 0-66 points; higher scores indicate better motor function and less impairment.
Time Frame: 60 days later
Population: All randomized participants completed the treatment and were included in the analysis. There were no dropouts or missing outcome data. The analysis was conducted on the full population according to the intention-to-treat principle.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group: Robot Rehand + Standard Rehabilitation | Control Group: Standard Rehabilitation Only
Number analyzed (Participants) | 60 | 60
score on a scale | 45.0 [42.0 to 49.0] | 36.0 [33.0 to 38.2]

2. Secondary Outcome: Barthel Index (BI)
Description: Barthel Index; range: 0-100 points; higher scores indicate greater independence in activities of daily living.
Time Frame: 60 days later
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group: Robot Rehand + Standard Rehabilitation | Control Group: Standard Rehabilitation Only
Number analyzed (Participants) | 60 | 60
score on a scale | 70.0 [68.8 to 70.0] | 55.0 [50.0 to 60.0]

3. Secondary Outcome: Functional Independence Measure Scale (FIM)
Description: Functional Independence Measure (FIM); range: 18-126 points; higher scores indicate greater functional independence.
Time Frame: 60 days later
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group: Robot Rehand + Standard Rehabilitation | Control Group: Standard Rehabilitation Only
Number analyzed (Participants) | 60 | 60
score on a scale | 76.0 [72.8 to 79.0] | 61.0 [59.0 to 63.0]

4. Secondary Outcome: National Institutes of Health Stroke Scale (NIHSS)
Description: National Institutes of Health Stroke Scale (NIHSS); range: 0-42 points; higher scores indicate more severe neurological impairment.
Time Frame: 60 days later
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group: Robot Rehand + Standard Rehabilitation | Control Group: Standard Rehabilitation Only
Number analyzed (Participants) | 60 | 60
score on a scale | 4.0 [2.0 to 7.0] | 6.5 [3.8 to 10.0]

5. Secondary Outcome: Frenchay Arm Test
Description: Frenchay Arm Test (FAT); range: 0-5 points; higher scores indicate better arm function.
Time Frame: 60 days later
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group: Robot Rehand + Standard Rehabilitation | Control Group: Standard Rehabilitation Only
Number analyzed (Participants) | 60 | 60
score on a scale | 3.0 [3.0 to 4.0] | 2.0 [1.0 to 2.0]

6. Secondary Outcome: Modified Wolf Motor Function Test (mWMFT)
Description: modified Wolf Motor Function Test (mWMFT); total score range: 0-75 points; higher scores indicate better upper extremity motor function.
Time Frame: 60 days later
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group: Robot Rehand + Standard Rehabilitation | Control Group: Standard Rehabilitation Only
Number analyzed (Participants) | 60 | 60
score on a scale | 53.0 [51.0 to 58.0] | 44.0 [42.0 to 46.2]

7. Secondary Outcome: Disabilities of the Arm Shoulder, and Hand (DASH) Test
Description: Disabilities of the Arm, Shoulder and Hand (DASH); range: 0-100 points; higher scores indicate greater disability.
Time Frame: 60 days later
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group: Robot Rehand + Standard Rehabilitation | Control Group: Standard Rehabilitation Only
Number analyzed (Participants) | 60 | 60
score on a scale | 17.0 [14.0 to 20.0] | 39.0 [35.8 to 41.0]

8. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: Hospital Anxiety and Depression Scale (HADS); range: 0-42 points; higher scores indicate greater psychological distress (more severe anxiety and depression symptoms).
Time Frame: 60 days later
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group: Robot Rehand + Standard Rehabilitation | Control Group: Standard Rehabilitation Only
Number analyzed (Participants) | 60 | 60
score on a scale | 16.0 [12.8 to 19.2] | 22.5 [19.0 to 26.0]

ADVERSE EVENTS:
Time Frame: From the first treatment session through the end of the 60-day intervention period.
Arm/Group | Intervention Group: Robot Rehand + Standard Rehabilitation | Control Group: Standard Rehabilitation Only
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 1/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group: Robot Rehand + Standard Rehabilitation (N=60) | Control Group: Standard Rehabilitation Only (N=60)
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT06937346/Prot_SAP_000.pdf